CLINICAL TRIAL: NCT05599815
Title: A Phase 2 Clinical Trial Investigating the Safety and Efficacy of ADX-629 in Subjects With Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome
Brief Title: Part 1 - A Clinical Trial in Patients With Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADX-629-MCD-001
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Nephrotic Syndrome
Keywords: Idiopathic nephrotic syndrome; Focal segmental glomerulosclerosis (FSGS); Minimal change disease; Frequently relapsing nephrotic syndrome; ADX-629; Reactive aldehyde species (RASP); Chronic kidney disease
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental; Renal Insufficiency, Chronic | interventions — ADX-629

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADX-629 (Experimental)
  Interventions: Drug: ADX-629

INTERVENTIONS:
Drug: ADX-629 — ADX-629 (250 milligrams) administered twice daily

SUMMARY:
A Clinical Trial Investigating the Safety and Efficacy of ADX-629 in Subjects with Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome

DETAILED DESCRIPTION:
ADX-629-MCD-001 is a multi-center, two-part, Phase 2 clinical trial designed to evaluate the safety and efficacy of ADX-629 in Subjects with frequently relapsing and steroid-dependent nephrotic syndrome. Study drug will be administered orally every 12 hours (twice daily) to eligible subjects for 90 days. The study will enroll approximately 35 children and adults with nephrotic syndrome who have had a nephrotic relapse in the 6 months prior to screening.

The clinical trial is divided into 2 parts: Part 1 (open-label) and Part 2 (double-blinded, randomized).

Part 1: Approximately 5 eligible subjects will receive open-label ADX-629 (250 mg) twice daily for 90 days.

Part 2: Approximately 30 eligible subjects will be randomized in a 2:1 ratio to receive either ADX-629 (250 mg) or matching placebo twice daily for 90 days.

Patients who are interested in participating will be provided detailed information about the study including description of study assessments/procedures, possible side-effects, alternative treatments, and potential benefits.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* History of nephrotic syndrome, characterized by heavy proteinuria and hypoalbuminemia
* Recent nephrotic relapse in the 6 months prior to screening
* Estimated glomerular filtration rate (eGFR) of ≥45 during screening
* Not pregnant, breastfeeding, or lactating and agree to use a highly effective method of acceptable contraceptive for the trial duration, if applicable

Exclusion Criteria:

* Subjects with collapsing FSGS focal segmental glomerulosclerosis (FSGS)
* Known secondary cause of nephrotic syndrome (e.g., diabetic nephropathy, systemic lupus erythematous, sickle cell anemia, malignancy, drug-induced, malaria)
* History of kidney transplantation or other solid organ transplantation
* History of any unstable chronic diseases/conditions, clinically significant abnormalities, or findings, that in the opinion of the Investigator, could compromise subject safety or affect the conduct of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) Query | From Day 1 to Day 90
  Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Relapse Frequency | From Day 1 to Day 90
  Proportion of subjects with one or more relapse(s), as defined by treatment with corticosteroid therapy

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Amicis Research Center - Northridge, Northridge, California
  - University of Colorado, Aurora, Colorado
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Emory University - Pediatric Nephrology, Atlanta, Georgia
  - ClinCept, LLC, Bremen, Georgia
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Nevada Kidney Disease Hypertension Center (NKDHC), Las Vegas, Nevada
  - East Carolina University - Nephrology, Greenville, North Carolina
  - The Ohio State University (OSU) Wexner Medical Center, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Southern Utah Kidney and Hypertension Center, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526